CLINICAL TRIAL: NCT01525615
Title: A Randomised, Double-blind, Placebo-controlled, Parallel Group Study to Determine the Effect of 12 Weeks Treatment of Orally Inhaled Tiotropium + Olodaterol Fixed Dose Combination (2.5/5 µg and 5/5 µg) Delivered by the Respimat® Inhaler, on Exercise Endurance Time During Constant Work Rate Cycle Ergometry in Patients With Chronic Obstructive Pulmonary Disease (COPD)[Torracto (TM)]
Brief Title: A Study to Determine the Effect of Tiotropium + Olodaterol Fixed Dose Combination on Exercise Endurance Time During Constant Work Rate Cycle Ergometry Test in COPD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1237.15; 2011-004253-11 (EudraCT Number: EudraCT)
Record Dates: First submitted 2012-02-01; First posted 2012-02-03 (Estimated); Results first posted 2015-09-15 (Estimated); Last update posted 2016-08-29 (Estimated); Status verified 2016-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — tiotropium-olodaterol; Tiotropium Bromide; olodaterol

ARMS (3):
- tiotropium+olodaterol low dose (Experimental): once daily 2 puffs, fixed dose combination (FDC) solution for inhalation Respimat
  Interventions: Device: Respimat inhaler; Drug: tiotropium+olodaterol (low dose)
- tiotropium+olodaterol high dose (Experimental): once daily 2 puffs, FDC solution for inhalation Respimat
  Interventions: Drug: tiotropium + olodaterol (high dose); Device: Respimat inhaler
- placebo (Placebo Comparator): once daily 2 puffs, solution for inhalation Respimat
  Interventions: Device: Respimat inhaler; Drug: placebo to tiotropium+olodaterol

INTERVENTIONS:
Device: Respimat inhaler — Respimat inhaler
  Arms: tiotropium+olodaterol low dose
Drug: tiotropium+olodaterol (low dose) — 2.5 µg tiotropium + 5 µg olodaterol
  Arms: tiotropium+olodaterol low dose
Drug: tiotropium + olodaterol (high dose) — 5 µg tiotropium + 5 µg olodaterol
  Arms: tiotropium+olodaterol high dose
Device: Respimat inhaler — Respimat inhaler
  Arms: tiotropium+olodaterol high dose
Device: Respimat inhaler — Respimat inhaler
  Arms: placebo
Drug: placebo to tiotropium+olodaterol — comparator
  Arms: placebo

SUMMARY:
The primary objective of this study is to compare the effects of orally inhaled tiotropium + olodaterol fixed dose combination (2.5/5 µg; 5/5 µg) with placebo on exercise tolerance after 12 weeks of treatment in patients with COPD.

ELIGIBILITY:
Inclusion criteria:

1. All patients must sign an informed consent consistent with ICH-GCP guidelines prior to participation in the trial, which includes medication washout and restrictions.
2. All patients must have a diagnosis of chronic obstructive pulmonary disease and must meet the following spirometric criteria:

   Patients must have relatively stable airway obstruction with, at visit 1:

   a post-bronchodilator 30% <= FEV1 <80% of predicted normal (ECSC) and a post-bronchodilator FEV1/FVC <70% at Visit 1
3. Male or female patients, between 40 and 75 years (inclusive) of age on day of signing informed consent.
4. Patients must be current or ex-smokers with a smoking history of more than 10 pack years Patients who have never smoked cigarettes must be excluded.
5. Patients must be able to perform technically acceptable pulmonary function tests (spirometry), must be able to complete multiple symptom-limited cycle ergometry tests (and for a subset also shuttle walk tests), as required in the protocol.
6. Patients must be able to inhale medication in a competent manner from the RESPIMAT inhaler and from a metered dose inhaler (MDI).

Exclusion criteria:

1. Patients with a significant disease other than COPD
2. Patients with clinically relevant abnormal baseline haematology, blood chemistry, or urinalysis; all patients with an SGOT > x2 ULN, SGPT > x2 ULN, bilirubin > x2 ULN or creatinine > x2 ULN will be excluded regardless of clinical condition
3. Patients with a history of asthma
4. A diagnosis of thyrotoxicosis
5. A diagnosis of paroxysmal tachycardia (>100 beats per minute)
6. A history of myocardial infarction within 1 year of screening visit (Visit 1)
7. Unstable or life-threatening cardiac arrhythmia
8. Hospitalized for heart failure within the past year
9. Known active tuberculosis
10. A malignancy for which patient has undergone resection, radiation therapy or chemotherapy within last five years
11. A history of life-threatening pulmonary obstruction and patients with chronic respiratory failure
12. A history of cystic fibrosis
13. Clinically evident bronchiectasis
14. A history of significant alcohol or drug abuse
15. Any contraindications for exercise testing
16. Patients who have undergone thoracotomy with pulmonary resection
17. Patients being treated with any oral ß-adrenergics
18. Patients being treated with oral corticosteroid medication at unstable doses (i.e., less than six weeks on a stable dose) or at doses in excess of the equivalent of 10 mg of prednisone per day or 20 mg every other day
19. Patients who regularly use daytime oxygen therapy for more than one hour per day and in the investigator's opinion will be unable to abstain from the use of oxygen therapy during clinic visits
20. Patients who have completed a pulmonary rehabilitation program in the six weeks prior to the screening visit (Visit 1) or patients who are currently in a pulmonary rehabilitation program
21. Patients who have a limitation of exercise performance as a result of factors other than fatigue or exertional dyspnoea or morbid obesity
22. Patients with an endurance time >=25 minutes during the training (Visit 2) or baseline (Visit 3) constant work rate cycle ergometry
23. Patients who have taken an investigational drug within one month or six half lives (whichever is greater) prior to screening visit (Visit 1)
24. Patients with known hypersensitivity to ß-adrenergic drugs, anticholinergic drugs, BAC, EDTA or any other component of the RESPIMAT inhalation solution delivery system
25. Pregnant or nursing women
26. Women of childbearing potential not using a highly effective method of birth control.

    Female patients will be considered to be of childbearing potential unless surgically sterilised by hysterectomy or bilateral tubal ligation, or post-menopausal for at least two years
27. Patients who have previously been randomized in this study or are currently participating in another study
28. Patients who are unable to comply with pulmonary medication restrictions prior to randomization

    At sites performing the shuttle walk tests, patients with the following criteria will be excluded from the shuttle walk tests:
29. Patients who complete level 12 at the incremental shuttle walk test at visit 1a.
30. Patients with an endurance time >=15 minutes during the training (Visit 2a) or baseline (visit 3a) endurance shuttle walk test.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 404 (Actual)
Dates: Start 2012-02; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (60):
- United States (15):
  - 1237.15.01503 Boehringer Ingelheim Investigational Site, Torrance, California
  - 1237.15.01512 Boehringer Ingelheim Investigational Site, Hartford, Connecticut
  - 1237.15.01506 Boehringer Ingelheim Investigational Site, Springfield, Illinois
  - 1237.15.01507 Boehringer Ingelheim Investigational Site, Iowa City, Iowa
  - 1237.15.01504 Boehringer Ingelheim Investigational Site, Livonia, Michigan
  - 1237.15.01511 Boehringer Ingelheim Investigational Site, Saint Charles, Missouri
  - 1237.15.01509 Boehringer Ingelheim Investigational Site, Lebanon, New Hampshire
  - 1237.15.01513 Boehringer Ingelheim Investigational Site, Charlotte, North Carolina
  - 1237.15.01514 Boehringer Ingelheim Investigational Site, Philadelphia, Pennsylvania
  - 1237.15.01516 Boehringer Ingelheim Investigational Site, Pittsburgh, Pennsylvania
  - 1237.15.01508 Boehringer Ingelheim Investigational Site, Easley, South Carolina
  - 1237.15.01501 Boehringer Ingelheim Investigational Site, Greenville, South Carolina
  - 1237.15.01505 Boehringer Ingelheim Investigational Site, Spartanburg, South Carolina
  - 1237.15.01502 Boehringer Ingelheim Investigational Site, Union, South Carolina
  - 1237.15.01510 Boehringer Ingelheim Investigational Site, Richmond, Virginia
- Argentina (3):
  - 1237.15.54502 Boehringer Ingelheim Investigational Site, Buenos Aires
  - 1237.15.54501 Boehringer Ingelheim Investigational Site, Mendonza
  - 1237.15.54503 Boehringer Ingelheim Investigational Site, Provincia de Buenos Aires
- Canada (5):
  - 1237.15.11501 Boehringer Ingelheim Investigational Site, Hamilotn, Ontario
  - 1237.15.11503 Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - 1237.15.11504 Boehringer Ingelheim Investigational Site, Kingston, Ontario
  - 1237.15.11505 Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - 1237.15.11502 Boehringer Ingelheim Investigational Site, Ste-Foy, Quebec
- Finland (3):
  - 1237.15.35851 Boehringer Ingelheim Investigational Site, Helsinki
  - 1237.15.35853 Boehringer Ingelheim Investigational Site, Turku
  - 1237.15.35852 Boehringer Ingelheim Investigational Site, Vaasa
- France (3):
  - 1237.15.33502 Boehringer Ingelheim Investigational Site, Nîmes
  - 1237.15.33504 Boehringer Ingelheim Investigational Site, Pessac
  - 1237.15.33501 Boehringer Ingelheim Investigational Site, Strasbourg
- Germany (8):
  - 1237.15.49507 Boehringer Ingelheim Investigational Site, Aschaffenburg
  - 1237.15.49502 Boehringer Ingelheim Investigational Site, Berlin
  - 1237.15.49504 Boehringer Ingelheim Investigational Site, Berlin
  - 1237.15.49501 Boehringer Ingelheim Investigational Site, Großhansdorf
  - 1237.15.49509 Boehringer Ingelheim Investigational Site, Hamburg
  - 1237.15.49505 Boehringer Ingelheim Investigational Site, Hanover
  - 1237.15.49508 Boehringer Ingelheim Investigational Site, Koblenz
  - 1237.15.49506 Boehringer Ingelheim Investigational Site, Wiesloch
- Hungary (4):
  - 1237.15.36504 Boehringer Ingelheim Investigational Site, Budapest
  - 1237.15.36501 Boehringer Ingelheim Investigational Site, Deszk
  - 1237.15.36503 Boehringer Ingelheim Investigational Site, Nyíregyháza
  - 1237.15.36502 Boehringer Ingelheim Investigational Site, Pécs
- Italy (8):
  - 1237.15.39512 Boehringer Ingelheim Investigational Site, Ferrara
  - 1237.15.39504 Boehringer Ingelheim Investigational Site, Parma
  - 1237.15.39503 Boehringer Ingelheim Investigational Site, Pavia
  - 1237.15.39501 Boehringer Ingelheim Investigational Site, Pisa
  - 1237.15.39509 Boehringer Ingelheim Investigational Site, Pisa
  - 1237.15.39511 Boehringer Ingelheim Investigational Site, Roma
  - 1237.15.39508 Boehringer Ingelheim Investigational Site, Sesto San Giovanni (MI)
  - 1237.15.39506 Boehringer Ingelheim Investigational Site, Trieste
- Spain (5):
  - 1237.15.34506 Boehringer Ingelheim Investigational Site, Alicante
  - 1237.15.34501 Boehringer Ingelheim Investigational Site, Barakaldo (Bilbao)
  - 1237.15.34507 Boehringer Ingelheim Investigational Site, Madrid
  - 1237.15.34009 Boehringer Ingelheim Investigational Site, Málaga
  - 1237.15.34001 Boehringer Ingelheim Investigational Site, Santander
- United Kingdom (6):
  - 1237.15.44152 Boehringer Ingelheim Investigational Site, Leicester
  - 1237.15.44154 Boehringer Ingelheim Investigational Site, Liverpool
  - 1237.15.44153 Boehringer Ingelheim Investigational Site, London
  - 1237.15.44151 Boehringer Ingelheim Investigational Site, Manchester
  - 1237.15.44155 Boehringer Ingelheim Investigational Site, Norwich
  - 1237.15.44158 Boehringer Ingelheim Investigational Site, Plymouth

REFERENCES:
- [Derived] Maltais F, O'Donnell D, Galdiz Iturri JB, Kirsten AM, Singh D, Hamilton A, Tetzlaff K, Zhao Y, Casaburi R. Effect of 12 weeks of once-daily tiotropium/olodaterol on exercise endurance during constant work-rate cycling and endurance shuttle walking in chronic obstructive pulmonary disease. Ther Adv Respir Dis. 2018 Jan-Dec;12:1753465818755091. doi: 10.1177/1753465818755091. PMID 29439648

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a randomised, placebo-controlled, double-blind, parallel-group comparison of once daily treatment with orally inhaled Tiotropium+Olodaterol Fixed Dose Combination (FDC) (2.5/5.0 µg; 5.0/5.0 µg) with placebo over 12 weeks.
Groups:
- Tio+Olo 2.5 / 5.0 µg: Oral inhalation of fixed dose combination (FDC) of Tiotropium 2.5 μg and Olodaterol 5 μg (Tiotropium: 1.25 μg per actuation and Olodaterol: 2.5 μg per actuation), 2 puffs from the RESPIMAT inhaler, once daily, in the morning.
- Tio+Olo 5.0 / 5.0 µg: Oral inhalation of FDC of Tiotropium 5 μg and Olodaterol 5 μg (Tiotropium and Olodaterol: 2.5 μg per actuation), 2 puffs from the RESPIMAT inhaler, once daily, in the morning.
Period: Overall Study
Arm/Group | Placebo | Tio+Olo 2.5 / 5.0 µg | Tio+Olo 5.0 / 5.0 µg
Started | 132 | 133 | 139
Completed | 118 | 126 | 133
Not Completed | 14 | 7 | 6
Not completed — Adverse Event | 11 | 7 | 5
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Other reason not described above | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Treated set included all randomised patients who were dispensed study medication and were documented to have taken any dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Tio+Olo 2.5 / 5.0 µg | Tio+Olo 5.0 / 5.0 µg | Total
Number analyzed (Participants) | 132 | 133 | 139 | 404
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (7.6) | 61.9 (7.3) | 63.1 (7.5) | 62.0 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 46 | 44 | 135
  Male | 87 | 87 | 95 | 269

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Mean Endurance Time During Constant Work Rate Cycle Ergometry (CWRCE) After 12 Weeks
Description: Primary endpoint was endurance time during constant work rate cycle ergometry to symptom limitation at 75% of maximal work capacity after 12 weeks of treatment. The endurance time in seconds was transformed using log10 scale to correct skewness in endurance time on original scale and then the MMRM model was fitted to the log10-transformed data and the least square means and SEs were obtained. To present the results in a way easier for interpretation, the least square mean from the MMRM fitted to the log10-transformed data were transformed back taking 10 to the power of the least square estimate for the log10 of geometric mean and the corresponding SE was transformed using delta method to get the corresponding SEs of the geometric mean.
Time Frame: 12 weeks
Population: Full analysis set (FAS). FAS is defined as all patients that were randomised, received treatment and had baseline and at least one post-baseline measurement before or at Week 12 for the primary endpoint.
Measure: Least Squares Mean (Standard Error); unit: seconds
Arm/Group | Placebo | Tio+Olo 2.5 / 5.0 µg | Tio+Olo 5.0 / 5.0 µg
Number analyzed (Participants) | 121 | 129 | 135
seconds | 463.63 (18.813) | 503.64 (19.642) | 527.51 (20.154)
Statistical Analysis 1: Comparison: Placebo vs Tio+Olo 5.0 / 5.0 µg; Treatment ratio between Tio+Olo 5.0/5.0 and placebo. This treatment comparison is the first one in the alpha-protected hierarchical testing chain; Test type: Superiority or Other; p = 0.0209, Mixed Models Analysis — Mixed effects Model for Repeated Measures (MMRM) with fixed effects of treatment, test day, treatment by test day interaction, log10 (baseline endurance time), log10 (baseline endurance time) by test day interaction, and patient as a random effect; Mean and 95% confidence limits were transformed from log10 back to the original scale. SE was calculated using the delta method; Treatment ratio = 1.138, 95% CI 2-sided [1.020 to 1.269], Standard Error of Mean 0.063
Statistical Analysis 2: Comparison: Placebo vs Tio+Olo 2.5 / 5.0 µg; Treatment ratio between Tio+Olo 2.5/5.0 and placebo. This treatment comparison is the second one in the alpha-protected hierarchical testing chain. Since the p-value for this treatment comparison is >0.05, the hierarchical testing chain is broken and all of the following hypothesis tests in this hierarchical chain are considered as descriptive only; Test type: Superiority or Other; p = 0.1419, Mixed Models Analysis — MMRM model for log10 (endurance time [s]) with fixed effects of treatment, test day, treatment by test day interaction, log10 (baseline endurance time [s]), log10 (baseline endurance time [s]) by test day interaction, patient as a random effect; [statistical method as in outcome 1, analysis 1]; Treatment ratio = 1.086, 95% CI 2-sided [0.973 to 1.213], Standard Error of Mean 0.061
Statistical Analysis 3: Comparison: Tio+Olo 2.5 / 5.0 µg vs Tio+Olo 5.0 / 5.0 µg; Treatment ratio between Tio+Olo 5.0/5.0 and Tio+Olo 2.5/5.0. This treatment comparison is not included in the alpha-protected hierarchical testing chain; Test type: Superiority or Other; p = 0.3970, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; [statistical method as in outcome 1, analysis 1]; Treatment ratio = 1.047, 95% CI 2-sided [0.941 to 1.166], Standard Error of Mean 0.057

2. Secondary Outcome: Adjusted Mean Endurance Time During Endurance Shuttle Walk Test (ESWT) After 12 Weeks
Description: Key secondary endpoint was endurance time during endurance shuttle walk test to symptom limitation at 85% of predicted maximum oxygen consumption (VO2) peak after 12 weeks of treatment. The endurance time in seconds was transformed using log10 scale to correct skewness in endurance time on original scale and then the MMRM model was fitted to the log10-transformed data and the least square means and SEs were obtained. To present the results in a way easier for interpretation, the least square mean from the MMRM fitted to the log10-transformed data were transformed back taking 10 to the power of the least square estimate for the log10 of geometric mean and the corresponding SE was transformed using delta method to get the corresponding SEs of the geometric mean.
Time Frame: 12 weeks
Population: Endurance shuttle walk test (ESWT) substudy set - This patient set included all patients in the Treated Set who had given informed consent for participating in the ESWT substudy and had a baseline and at least one post-baseline measurement during ESWT before or at Week 12 for the key secondary endpoint.
Measure: Least Squares Mean (Standard Error); unit: seconds
Arm/Group | Placebo | Tio+Olo 2.5 / 5.0 µg | Tio+Olo 5.0 / 5.0 µg
Number analyzed (Participants) | 50 | 56 | 59
seconds | 311.41 (22.519) | 377.20 (25.942) | 376.39 (25.033)
Statistical Analysis 1: Comparison: Placebo vs Tio+Olo 5.0 / 5.0 µg; Treatment ratio between Tio+Olo 5.0/5.0 and placebo. Since the hierarchical testing chain has been broken, even though this treatment comparison is included as the 3rd one in the alpha-protected hierarchical testing chain, this hypothesis test is descriptive only; Test type: Superiority or Other; p = 0.0552, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; [statistical method as in outcome 1, analysis 1]; Tretament ratio = 1.209, 95% CI 2-sided [0.996 to 1.467], Standard Error of Mean 0.119
Statistical Analysis 2: Comparison: Placebo vs Tio+Olo 2.5 / 5.0 µg; Treatment ratio between Tio+Olo 2.5/5.0 and placebo; Test type: Superiority or Other; p = 0.0562, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; Mean, 95% confidence limits transformed from log10 to original scale. SE was calculated using the delta method. This hypothesis test is descriptive; Treatment ratio = 1.211, 95% CI 2-sided [0.995 to 1.475], Standard Error of Mean 0.121
Statistical Analysis 3: Comparison: Tio+Olo 2.5 / 5.0 µg vs Tio+Olo 5.0 / 5.0 µg; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.9822, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; [statistical method as in outcome 1, analysis 1]; Treatment ratio = 0.998, 95% CI 2-sided [0.826 to 1.205], Standard Error of Mean 0.095

3. Secondary Outcome: Adjusted Mean Inspiratory Capacity at Pre-exercise After 12 Weeks
Description: Secondary endpoint was pre-exercise inspiratory capacity (IC) before constant work rate cycle ergometry to symptom limitation at 75% maximal work capacity (Wcap) after 12 weeks of treatment.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Tio+Olo 2.5 / 5.0 µg | Tio+Olo 5.0 / 5.0 µg
Number analyzed (Participants) | 119 | 128 | 133
liters | 2.390 (0.038) | 2.597 (0.036) | 2.624 (0.035)
Statistical Analysis 1: Comparison: Placebo vs Tio+Olo 5.0 / 5.0 µg; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — MMRM model for inspiratory capacity with fixed effects of treatment, test day, treatment by test day interaction, baseline inspiratory capacity, baseline inspiratory capacity by test day interaction, and patient as a random effect; This hypothesis test is descriptive; LSMean Difference-Final Values = 0.234, 95% CI 2-sided [0.133 to 0.336], Standard Error of Mean 0.052 — LSMean=Least square mean
Statistical Analysis 2: Comparison: Placebo vs Tio+Olo 2.5 / 5.0 µg; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; This hypothesis test is descriptive; LSMean Difference-Final Values = 0.207, 95% CI 2-sided [0.105 to 0.309], Standard Error of Mean 0.052
Statistical Analysis 3: Comparison: Tio+Olo 2.5 / 5.0 µg vs Tio+Olo 5.0 / 5.0 µg; Test type: Superiority or Other; p = 0.5892, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; This hypothesis test is descriptive; LSMean Difference-Final Values = 0.027, 95% CI 2-sided [-0.072 to 0.126], Standard Error of Mean 0.050

4. Secondary Outcome: Adjusted Mean Endurance Time During Constant Work Rate Cycle Ergometry (CWRCE) on Day 1
Description: Secondary endpoint was endurance time during constant work rate cycle ergometry to symptom limitation at 75% of maximal work capacity on Day 1. Analysis of covariance model on log10 transformation data. Adjusted means are back transformed to report in original units. Standard errors (SEs) are calculated using the delta method.
Time Frame: 1 day
Population: Visit 4 Set. All randomized patients dispensed medication, were documented to have taken any dose of study medication, and had evaluable measurements of endurance time at Baseline (Visit 3) and at Visit 4 (Day 1) during CWRCE. Patients were assigned to the Visit 4 set after implementation of data handling rules that set measurements to missing.
Measure: Least Squares Mean (Standard Error); unit: seconds
Arm/Group | Placebo | Tio+Olo 2.5 / 5.0 µg | Tio+Olo 5.0 / 5.0 µg
Number analyzed (Participants) | 77 | 77 | 80
seconds | 478.59 (17.861) | 527.69 (19.670) | 538.76 (19.715)
Statistical Analysis 1: Comparison: Placebo vs Tio+Olo 5.0 / 5.0 µg; Treatment ratio between Tio+Olo 5.0/5.0 and placebo; Test type: Superiority or Other; p = 0.0245, ANCOVA — ANCOVA model for log10 (endurance time [s]) with categorical effects of treatment and (log10-transformed) baseline as continuous covariate; This hypothesis test is descriptive; Treatment ratio = 1.126, 95% CI 2-sided [1.015 to 1.248], Standard Error of Mean 0.059
Statistical Analysis 2: Comparison: Placebo vs Tio+Olo 2.5 / 5.0 µg; Treatment ratio between Tio+Olo 2.5/5.0 and placebo; Test type: Superiority or Other; p = 0.0655, ANCOVA; Descriptive; Treatment ratio = 1.103, 95% CI 2-sided [0.994 to 1.223], Standard Error of Mean 0.058
Statistical Analysis 3: Comparison: Tio+Olo 2.5 / 5.0 µg vs Tio+Olo 5.0 / 5.0 µg; Treatment ratio between Tio+Olo 5.0/5.0 and Tio+Olo 2.5/5.0; Test type: Superiority or Other; p = 0.6912, ANCOVA; Descriptive; Treatment ratio = 1.021, 95% CI 2-sided [0.921 to 1.132], Standard Error of Mean 0.053

5. Secondary Outcome: Adjusted Mean Endurance Time During Constant Work Rate Cycle Ergometry (CWRCE) After 6 Weeks Treatment
Description: Secondary endpoint was endurance time during constant work rate cycle ergometry to symptom limitation at 75% of maximal work capacity after 6 weeks of treatment.The endurance time in seconds was transformed using log10 scale to correct skewness in endurance time on original scale and then the MMRM model was fitted to the log10-transformed data and the least square means and SEs were obtained. To present the results in a way easier for interpretation, the least square mean from the MMRM fitted to the log10-transformed data were transformed back taking 10 to the power of the least square estimate for the log10 of geometric mean and the corresponding SE was transformed using delta method to get the corresponding SEs of the geometric mean.
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: seconds
Arm/Group | Placebo | Tio+Olo 2.5 / 5.0 µg | Tio+Olo 5.0 / 5.0 µg
Number analyzed (Participants) | 121 | 129 | 135
seconds | 427.74 (17.093) | 522.26 (20.232) | 525.62 (19.990)
Statistical Analysis 1: Comparison: Placebo vs Tio+Olo 5.0 / 5.0 µg; Treatment ratio between Tio+Olo 5.0/5.0 and placebo. Hypothesis test is descriptive; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; [statistical method as in outcome 1, analysis 1]; Treatment ratio = 1.229, 95% CI 2-sided [1.103 to 1.370], Standard Error of Mean 0.068
Statistical Analysis 2: Comparison: Placebo vs Tio+Olo 2.5 / 5.0 µg; Treatment ratio between Tio+Olo 2.5/5.0 and placebo. Hypothesis test is descriptive; Test type: Superiority or Other; p = 0.0004, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; [statistical method as in outcome 1, analysis 1]; Treatment ratio = 1.221, 95% CI 2-sided [1.095 to 1.362], Standard Error of Mean 0.068
Statistical Analysis 3: Comparison: Tio+Olo 2.5 / 5.0 µg vs Tio+Olo 5.0 / 5.0 µg; Treatment ratio between Tio+Olo 5.0/5.0 and Tio+Olo 2.5/5.0. Hypothesis test is descriptive; Test type: Superiority or Other; p = 0.9062, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; [statistical method as in outcome 1, analysis 1]; Treatment ratio = 1.006, 95% CI 2-sided [0.905 to 1.12], Standard Error of Mean 0.055

6. Secondary Outcome: Adjusted Mean Inspiratory Capacity at Pre-exercise After 1 Day
Description: Secondary endpoint was pre-exercise inspiratory capacity (IC) during constant work rate cycle ergometry to symptom limitation at 75% maximal work capacity (Wcap) on Day 1.
Time Frame: 1 day
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Tio+Olo 2.5 / 5.0 µg | Tio+Olo 5.0 / 5.0 µg
Number analyzed (Participants) | 75 | 77 | 76
liters | 2.440 (0.041) | 2.642 (0.041) | 2.605 (0.041)
Statistical Analysis 1: Comparison: Placebo vs Tio+Olo 5.0 / 5.0 µg; Test type: Superiority or Other; p = 0.0049, ANCOVA — ANCOVA model for inspiratory capacity (liters) with categorical effect of treatment and baseline as continuous covariate; Descriptive; LSMean Difference-Final Values = 0.165, 95% CI 2-sided [0.051 to 0.279], Standard Error of Mean 0.058
Statistical Analysis 2: Comparison: Placebo vs Tio+Olo 2.5 / 5.0 µg; Test type: Superiority or Other; p = 0.0006, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Descriptive; LSMean Difference-Final Values = 0.202, 95% CI 2-sided [0.088 to 0.316], Standard Error of Mean 0.058
Statistical Analysis 3: Comparison: Tio+Olo 2.5 / 5.0 µg vs Tio+Olo 5.0 / 5.0 µg; Test type: Superiority or Other; p = 0.5162, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Descriptive; LSMean Difference-Final Values = -0.037, 95% CI 2-sided [-0.151 to 0.076], Standard Error of Mean 0.058

7. Secondary Outcome: Adjusted Mean Inspiratory Capacity at Pre-exercise After 6 Weeks
Description: Secondary endpoint was pre-exercise inspiratory capacity (IC) during constant work rate cycle ergometry to symptom limitation at 75% maximal work capacity (Wcap) after 6 weeks of treatment.
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Tio+Olo 2.5 / 5.0 µg | Tio+Olo 5.0 / 5.0 µg
Number analyzed (Participants) | 119 | 128 | 133
liters | 2.402 (0.037) | 2.589 (0.036) | 2.627 (0.035)
Statistical Analysis 1: Comparison: Placebo vs Tio+Olo 5.0 / 5.0 µg; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; Descriptive; LSMean Difference-Final Values = 0.225, 95% CI 2-sided [0.124 to 0.326], Standard Error of Mean 0.051
Statistical Analysis 2: Comparison: Placebo vs Tio+Olo 2.5 / 5.0 µg; Test type: Superiority or Other; p = 0.0003, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; Descriptive; LSMean Difference-Final Values = 0.187, 95% CI 2-sided [0.086 to 0.288], Standard Error of Mean 0.052
Statistical Analysis 3: Comparison: Tio+Olo 2.5 / 5.0 µg vs Tio+Olo 5.0 / 5.0 µg; Test type: Superiority or Other; p = 0.4541, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; Descriptive; LSMean Difference-Final Values = 0.038, 95% CI 2-sided [-0.061 to 0.137], Standard Error of Mean 0.050

8. Secondary Outcome: Adjusted Mean Slope of the Intensity of Breathing Discomfort on Day 1
Description: Secondary endpoint was the slope of the intensity of breathing discomfort during constant work rate cycle ergometry to symptom limitation at 75% of maximal work capacity after 1 day of treatment.
  The intensity of breathing discomfort was rated on the Borg Scale with categories from 0 (nothing at all) to 10 (maximal). The slope of the intensity of breathing discomfort was defined as the Borg scale value of breathing discomfort at the end of exercise minus the Borg scale value of breathing discomfort at pre-exercise divided by the endurance time. A decrease in slope indicates slowing down in decline in breathing, i.e., favorable results.
Time Frame: 1 day
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: units / seconds
Arm/Group | Placebo | Tio+Olo 2.5 / 5.0 µg | Tio+Olo 5.0 / 5.0 µg
Number analyzed (Participants) | 76 | 77 | 80
units / seconds | 0.014 (0.001) | 0.012 (0.001) | 0.012 (0.001)
Statistical Analysis 1: Comparison: Placebo vs Tio+Olo 5.0 / 5.0 µg; Test type: Superiority or Other; p = 0.0468, ANCOVA — ANCOVA model for mean slope of the intensity of breathing discomfort with categorical effect of treatment and baseline as continuous covariate; Descriptive; LSMean Difference-Final Values = -0.002, 95% CI 2-sided [-0.004 to -0.000], Standard Error of Mean 0.001
Statistical Analysis 2: Comparison: Placebo vs Tio+Olo 2.5 / 5.0 µg; Test type: Superiority or Other; p = 0.0180, ANCOVA — [p-value comment as in outcome 8, analysis 1]; Descriptive; LSMean Difference-Final Values = -0.002, 95% CI 2-sided [-0.005 to -0.000], Standard Error of Mean 0.001
Statistical Analysis 3: Comparison: Tio+Olo 2.5 / 5.0 µg vs Tio+Olo 5.0 / 5.0 µg; Test type: Superiority or Other; p = 0.6856, ANCOVA — [p-value comment as in outcome 8, analysis 1]; Descriptive; LSMean Difference-Final Values = 0.000, 95% CI 2-sided [-0.002 to 0.002], Standard Error of Mean 0.001

9. Secondary Outcome: Adjusted Mean Slope of the Intensity of Breathing Discomfort After Week 6
Description: Secondary endpoint was the slope of the intensity of breathing discomfort during constant work rate cycle ergometry to symptom limitation at 75% of maximal work capacity after 6 weeks of treatment.
  The intensity of breathing discomfort was rated on the Borg Scale with categories from 0 (nothing at all) to 10 (maximal). The slope of the intensity of breathing discomfort was defined as the Borg scale value of breathing discomfort at the end of exercise minus the Borg scale value of breathing discomfort at pre-exercise divided by the endurance time. A decrease in slope indicates favorable results.
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units / seconds
Arm/Group | Placebo | Tio+Olo 2.5 / 5.0 µg | Tio+Olo 5.0 / 5.0 µg
Number analyzed (Participants) | 120 | 129 | 135
units / seconds | 0.016 (0.001) | 0.013 (0.001) | 0.013 (0.001)
Statistical Analysis 1: Comparison: Placebo vs Tio+Olo 5.0 / 5.0 µg; Test type: Superiority or Other; p = 0.0081, Mixed Models Analysis — MMRM model with fixed effects of treatment, test day, treatment by test day interaction, baseline, baseline by test day interaction, and patient as a random effect; Descriptive; LSMean Difference-Final Values = -0.003, 95% CI 2-sided [-0.005 to -0.001], Standard Error of Mean 0.001
Statistical Analysis 2: Comparison: Placebo vs Tio+Olo 2.5 / 5.0 µg; Test type: Superiority or Other; p = 0.0099, Mixed Models Analysis — [p-value comment as in outcome 9, analysis 1]; Descriptive; LSMean Difference-Final Values = -0.003, 95% CI 2-sided [-0.005 to -0.001], Standard Error of Mean 0.001
Statistical Analysis 3: Comparison: Tio+Olo 2.5 / 5.0 µg vs Tio+Olo 5.0 / 5.0 µg; Test type: Superiority or Other; p = 0.9626, Mixed Models Analysis — [p-value comment as in outcome 9, analysis 1]; Descriptive; LSMean Difference-Final Values = -0.000, 95% CI 2-sided [-0.002 to 0.002], Standard Error of Mean 0.001

10. Secondary Outcome: Adjusted Mean Slope of the Intensity of Breathing Discomfort After Week 12
Description: Secondary endpoint was the slope of the intensity of breathing discomfort during constant work rate cycle ergometry to symptom limitation at 75% of maximal work capacity after 12 weeks of treatment.
  The intensity of breathing discomfort was rated on the Borg Scale with categories from 0 (nothing at all) to 10 (maximal). The slope of the intensity of breathing discomfort was defined as the Borg scale value of breathing discomfort at the end of exercise minus the Borg scale value of breathing discomfort at pre-exercise divided by the endurance time. A decrease in slope indicates favorable results.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units / seconds
Arm/Group | Placebo | Tio+Olo 2.5 / 5.0 µg | Tio+Olo 5.0 / 5.0 µg
Number analyzed (Participants) | 120 | 129 | 135
units / seconds | 0.015 (0.001) | 0.013 (0.001) | 0.013 (0.001)
Statistical Analysis 1: Comparison: Placebo vs Tio+Olo 5.0 / 5.0 µg; Test type: Superiority or Other; p = 0.0598, Mixed Models Analysis — [p-value comment as in outcome 9, analysis 1]; Descriptive; LSMean Difference-Final Values = -0.002, 95% CI 2-sided [-0.004 to 0.000], Standard Error of Mean 0.001
Statistical Analysis 2: Comparison: Placebo vs Tio+Olo 2.5 / 5.0 µg; Test type: Superiority or Other; p = 0.0218, Mixed Models Analysis — [p-value comment as in outcome 9, analysis 1]; Descriptive; LSMean Difference-Final Values = -0.003, 95% CI 2-sided [-0.005 to -0.000], Standard Error of Mean 0.001
Statistical Analysis 3: Comparison: Tio+Olo 2.5 / 5.0 µg vs Tio+Olo 5.0 / 5.0 µg; Test type: Superiority or Other; p = 0.6549, Mixed Models Analysis — [p-value comment as in outcome 9, analysis 1]; Descriptive; LSMean Difference-Final Values = 0.000, 95% CI 2-sided [-0.002 to 0.003], Standard Error of Mean 0.001

11. Secondary Outcome: Adjusted Mean 1-hour, Post-dose Forced Expiratory Volume in One Second (FEV1) on Day 1
Description: Secondary endpoint was adjusted mean 1-hour, post-dose Forced Expiratory Volume in one second (FEV1) observed on day 1
Time Frame: 1 day
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Tio+Olo 2.5 / 5.0 µg | Tio+Olo 5.0 / 5.0 µg
Number analyzed (Participants) | 121 | 129 | 135
liters | 1.509 (0.020) | 1.693 (0.019) | 1.679 (0.019)
Statistical Analysis 1: Comparison: Placebo vs Tio+Olo 5.0 / 5.0 µg; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 9, analysis 1]; Descriptive; LSMean Difference-Final Values = 0.170, 95% CI 2-sided [0.116 to 0.224], Standard Error of Mean 0.028
Statistical Analysis 2: Comparison: Placebo vs Tio+Olo 2.5 / 5.0 µg; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 9, analysis 1]; Descriptive; LSMean Difference-Final Values = 0.184, 95% CI 2-sided [0.129 to 0.239], Standard Error of Mean 0.028
Statistical Analysis 3: Comparison: Tio+Olo 2.5 / 5.0 µg vs Tio+Olo 5.0 / 5.0 µg; Test type: Superiority or Other; p = 0.6105, Mixed Models Analysis — [p-value comment as in outcome 9, analysis 1]; Descriptive; LSMean Difference-Final Values = -0.014, 95% CI 2-sided [-0.067 to 0.040], Standard Error of Mean 0.027

12. Secondary Outcome: Adjusted Mean 1-hour, Post-dose Forced Expiratory Volume in One Second (FEV1) After 6 Weeks
Description: Secondary endpoint was adjusted mean 1-hour, post-dose Forced Expiratory Volume in one second (FEV1) observed after 6 weeks of treatment
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Tio+Olo 2.5 / 5.0 µg | Tio+Olo 5.0 / 5.0 µg
Number analyzed (Participants) | 121 | 129 | 135
liters | 1.517 (0.020) | 1.790 (0.019) | 1.763 (0.019)
Statistical Analysis 1: Comparison: Placebo vs Tio+Olo 5.0 / 5.0 µg; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 9, analysis 1]; Descriptive; LSMean Difference-Final Values = 0.246, 95% CI 2-sided [0.192 to 0.300], Standard Error of Mean 0.028
Statistical Analysis 2: Comparison: Placebo vs Tio+Olo 2.5 / 5.0 µg; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 9, analysis 1]; Descriptive; LSMean Difference-Final Values = 0.273, 95% CI 2-sided [0.218 to 0.328], Standard Error of Mean 0.028
Statistical Analysis 3: Comparison: Tio+Olo 2.5 / 5.0 µg vs Tio+Olo 5.0 / 5.0 µg; Test type: Superiority or Other; p = 0.3236, Mixed Models Analysis — [p-value comment as in outcome 9, analysis 1]; Descriptive; LSMean Difference-Final Values = -0.027, 95% CI 2-sided [-0.080 to 0.027], Standard Error of Mean 0.027

13. Secondary Outcome: Adjusted Mean 1-hour, Post-dose Forced Expiratory Volume in One Second (FEV1) After 12 Weeks
Description: Secondary endpoint was adjusted mean 1-hour, post-dose Forced Expiratory Volume in one second (FEV1) observed after 12 weeks of treatment
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Tio+Olo 2.5 / 5.0 µg | Tio+Olo 5.0 / 5.0 µg
Number analyzed (Participants) | 121 | 129 | 135
liters | 1.527 (0.020) | 1.784 (0.019) | 1.778 (0.019)
Statistical Analysis 1: Comparison: Placebo vs Tio+Olo 5.0 / 5.0 µg; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 9, analysis 1]; Descriptive; LSMean Difference-Final Values = 0.251, 95% CI 2-sided [0.196 to 0.305], Standard Error of Mean 0.028
Statistical Analysis 2: Comparison: Placebo vs Tio+Olo 2.5 / 5.0 µg; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 9, analysis 1]; Descriptive; LSMean Difference-Final Values = 0.257, 95% CI 2-sided [0.202 to 0.312], Standard Error of Mean 0.028
Statistical Analysis 3: Comparison: Tio+Olo 2.5 / 5.0 µg vs Tio+Olo 5.0 / 5.0 µg; Test type: Superiority or Other; p = 0.8156, Mixed Models Analysis — [p-value comment as in outcome 9, analysis 1]; Descriptive; LSMean Difference-Final Values = -0.006, 95% CI 2-sided [-0.060 to 0.047], Standard Error of Mean 0.027

ADVERSE EVENTS:
Time Frame: 142 days
Description: All adverse events, occurring during the course of the clinical trial (i.e. from signing the informed consent onwards throughout the 12 week treatment period and the 21-day follow up period) were to be collected, documented, and reported to the sponsor on the appropriate electronic case report form / serious adverse event reporting forms.
Groups:
- Placebo: once daily 2 puffs, solution for inhalation Respimat placebo to tiotropium+olodaterol: comparator
- Tio+Olo 2.5 / 5.0 μg: Oral inhalation of fixed dose combination (FDC) of Tiotropium 2.5 μg and Olodaterol 5 μg (Tiotropium: 1.25 μg per actuation and Olodaterol: 2.5 μg per actuation), 2 puffs from the RESPIMAT inhaler, once daily, in the morning.
- Tio+Olo 5.0 / 5.0 μg: Oral inhalation of FDC of Tiotropium 5 μg and Olodaterol 5 μg (Tiotropium and Olodaterol: 2.5 μg per actuation), 2 puffs from the RESPIMAT inhaler, once daily, in the morning.
Arm/Group | Placebo | Tio+Olo 2.5 / 5.0 μg | Tio+Olo 5.0 / 5.0 μg
Serious Adverse Events (participants affected / at risk) | 5/132 | 9/133 | 4/139
Other Adverse Events (participants affected / at risk) | 25/132 | 25/133 | 16/139
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=132) | Tio+Olo 2.5 / 5.0 μg (N=133) | Tio+Olo 5.0 / 5.0 μg (N=139)
Angina pectoris (Cardiac disorders) | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastases to adrenals (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=132) | Tio+Olo 2.5 / 5.0 μg (N=133) | Tio+Olo 5.0 / 5.0 μg (N=139)
Nasopharyngitis (Infections and infestations) | 6 | 9 | 4
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 15 | 10 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 9 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.